CLINICAL TRIAL: NCT02402465
Title: Evaluating Factors Involved in Dymista's Superior Clinical Efficacy to Fluticasone Propionate in the Treatment of Seasonal Allergic Rhinitis
Brief Title: Factors Involved in Dymista's Superior Clinical Efficacy in the Treatment of Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB14-1199
Record Dates: First submitted 2015-03-18; First posted 2015-03-30 (Estimated); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-02

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Sodium Chloride; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo nasal spray that is similar to Dymista in all respects except the active ingredient
  Interventions: Drug: Placebo; Procedure: Nasal Allergen Challenge
- Fluticasone propionate (Experimental): Fluticasone propionate nasal spray provided in a bottle similar to placebo and dymista
  Interventions: Drug: Fluticasone propionate; Procedure: Nasal Allergen Challenge
- Dymista (fluticasone/azelastine) (Experimental): Dymista is also provided as a nasal spray in bottles similar to the other two agents
  Interventions: Drug: Fluticasone/Azelastine nasal spray; Procedure: Nasal Allergen Challenge

INTERVENTIONS:
Drug: Placebo — Patients will be treated by placebo
  Other Names: saline
  Arms: Placebo
Drug: Fluticasone propionate — Patients will receive fluticasone nasal spray
  Other Names: Flonase
  Arms: Fluticasone propionate
Drug: Fluticasone/Azelastine nasal spray — Patients will receive Dymista nasal spray
  Other Names: Dymista
  Arms: Dymista (fluticasone/azelastine)
Procedure: Nasal Allergen Challenge — All subjects will receive a nasal challenge with allergen to mimick an allergic response and allow the investigation of the different drug effects on that response. Allergen extracts will be used as sprays into the nasal cavity. The extracts are approved by FDA for skin testing or desensitization therapy and an IND was obtained to allow intranasal administration
  Other Names: Nasal provocation

SUMMARY:
Dymista, a combined product containing the antihistamine azelastine and the intranasal steroid fluticasone, provides superior clinical efficacy to both fluticasone propionate and azelastine hydrochloride in the treatment of seasonal allergic rhinitis. The superiority of efficacy not only occurs at the initiation of treatment, but persists for its duration. The mechanism underlying the superior efficacy of Dymista is not known. This trial focuses on examining the effects of Dymista on the dynamics of the allergic response in man using nasal provocation with antigen. The investigators will study the relationship between symptoms, physiology, cells and mediators.

DETAILED DESCRIPTION:
The main hypothesis for the trial is that Dymista affects multiple phases of the allergic response, which in sum are greater than the effects of fluticasone propionate or azelastine hydrochloride alone.

Our objectives for this study are to demonstrate:

1. that the induction of allergic inflammation by nasal provocation with antigen causes a cellular infiltration, with subsequent release of inflammatory biomarkers that cause augmented responses to subsequent exposure to antigens.
2. that fluticasone prevents allergic inflammation from developing after antigen challenge and subsequently prevents the augmentation of the nasal response to nasal challenge with antigen.
3. that the azelastine in Dymista reduces the effects of released histamine

To address these hypotheses we will perform a 3-way, randomized, placebo-controlled, and crossover trial. We will recruit 20 asymptomatic seasonal allergic rhinitis patients outside of the relevant season. The subjects will receive placebo, fluticasone propionate and Dymista. The nasal provocations will be separated by 2 weeks. Treatment will begin 15 minutes before nasal provocation with ragweed or grass antigen and the treatment will continue twice a day for 3 days. Nasal provocation will occur daily for three days to evaluate for priming (increased sensitization with repeated antigen exposure, which mimics seasonal disease where antigen exposure occurs in the setting of continued allergic inflammation). For outcome measures, we will monitor both nasal symptoms after nasal provocation as well as collect nasal lavage to evaluate effects on eosinophils and biomarkers of the immune response. In the nasal lavage, we will quantify the number of eosinophils (a marker of cellular recruitment) and measure the levels of histamine (a marker of basophil and mast cell activation), tryptase (a marker of mast cell activation), albumin (a marker of vascular permeability), lactoferrin (a marker of glandular activation) and ECP (a marker of eosinophil activation). Thus we expect to generate information on both clinical effects and physiologic differences between the treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 18 and 55 years of age.
2. History of grass and/or ragweed allergic rhinitis.
3. Positive skin test to grass and/or ragweed antigen.
4. Positive response to screening nasal challenge.
5. Off all anti-allergic medications for a minimum of 2 weeks.

Exclusion Criteria:

1. Physical signs or symptoms suggestive of renal, hepatic or cardiovascular disease.
2. Pregnant or lactating women.
3. Upper respiratory infection within 14 days of study start.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2020-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fuad M Baroody, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago Medicine, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: cross-over study
Groups:
- Dymista/Placebo/Flonase: Randomized order of Dymista, then Placebo, then Flonase
- Dymista/Flonase/Placebo: Randomized order of Dymista, then Flonase, then Placebo
- Placebo/Dymista/Flonase: Randomized order of Placebo, then Dymista, then Flonase
- Placebo/Flonase/Dymista: Randomized order of Placebo, then Flonase, then Dymista
- Flonase/Dymista/Placebo: Randomized order of Flonase, then Dymista, then Placebo
- Flonase/Placebo/Dymista: Randomized order of Flonase, then Placebo, then Dymista
Period: Overall Study
Arm/Group | Dymista/Placebo/Flonase | Dymista/Flonase/Placebo | Placebo/Dymista/Flonase | Placebo/Flonase/Dymista | Flonase/Dymista/Placebo | Flonase/Placebo/Dymista
Started | 4 | 4 | 4 | 4 | 2 | 4
Completed | 4 | 3 | 4 | 4 | 1 | 3
Not Completed | 0 | 1 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: This is a cross-over study.
Groups:
- Dymista/Placebo/Flonase; Dymista/Flonase/Placebo; Placebo/Dymista/Flonase; Placebo/Flonase/Dymista; Flonase/Dymista/Placebo; Flonase/Placebo/Dymista: Dymista:
  Fluticasone/Azelastine nasal spray
  Flonase: Fluticasone nasal spray
  Placebo: nasal spray without active ingredient
- Total: Total of all reporting groups
Arm/Group | Dymista/Placebo/Flonase | Dymista/Flonase/Placebo | Placebo/Dymista/Flonase | Placebo/Flonase/Dymista | Flonase/Dymista/Placebo | Flonase/Placebo/Dymista | Total
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 1 | 3 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 4 | 4 | 1 | 3 | 19
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 34.5 [21 to 46] | 29 [21 to 54] | 29 [21 to 43] | 27 [18 to 46] | 42 [42 to 42] | 36 [35 to 52] | 34 [18 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 3 | 1 | 0 | 2 | 10
  Male | 3 | 0 | 1 | 3 | 1 | 1 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 1 | 0 | 0 | 3
  Not Hispanic or Latino | 3 | 2 | 4 | 3 | 1 | 3 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 2 | 2 | 1 | 3 | 11
  White | 1 | 1 | 2 | 1 | 0 | 0 | 5
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 1 | 0 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 4 | 4 | 1 | 3 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Response in Albumin Levels in Nasal Lavage Following Each Challenge
Description: Our procedure used a diluent (sham) challenge followed by 2 allergen challenges where lavages are collected 10 minutes after each of these challenges. The final value is (albumin amount in lavage after 1st allergen exposure - amount after sham) + (amount in lavage after 2nd exposure - sham amount).
Time Frame: 3 rounds of 1 Nasal challenge every 3 days followed by 2 week washout periods in between. Total participation of 9 weeks.
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Fluticasone Propionate | Dymista (Fluticasone/Azelastine)
Number analyzed (Participants) | 19 | 19 | 19
ng/mL
  day 1 | -33.61 (53.03) | -82.2 (54.22) | -185.85 (158.04)
  day 2 | -41.87 (59.22) | -29.70 (72.14) | -81.6 (32.36)
  day 3 | -106.68 (46.08) | -78.73 (58.44) | -69.50 (35.49)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Propionate vs Dymista (Fluticasone/Azelastine); Test type: Superiority; p > 0.05, ANOVA; Mean Difference (Final Values) = 37 — Mean difference is related to albumin levels in nasal lavages: Unit= ng/ml

2. Secondary Outcome: Sneezes After Allergen Challenge
Description: Our procedure used a diluent (sham) challenge followed by 2 allergen challenges. The final value is (the number of sneezes after 1st allergen exposure - number after sham) + (number of sneezes after 2nd exposure - sham amount).
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: Sneezes
Arm/Group | Placebo | Fluticasone Propionate | Dymista (Fluticasone/Azelastine)
Number analyzed (Participants) | 19 | 19 | 19
Sneezes
  day 1 | 6.2 (2.2) | 6.8 (1.6) | 1.1 (0.5)
  Day 2 | 9.3 (2.6) | 7.6 (2.2) | 2.0 (0.9)
  day 3 | 9.0 (2.5) | 7.1 (2.0) | 2.1 (0.9)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Propionate vs Dymista (Fluticasone/Azelastine); Test type: Superiority; p = 0.001, Friedman — Bonferroni correction was used to adjust for the fact that each day was tested separately yielding alpha=0.05/3; Non-parametric repeated measures ANOVA; Friedman's Q = 14.2
Statistical Analysis 2: Comparison: Placebo vs Dymista (Fluticasone/Azelastine); Test type: Superiority; p = 0.02, Wilcoxon (Mann-Whitney); Median Difference (Net) = 24.5
Statistical Analysis 3: Comparison: Fluticasone Propionate vs Dymista (Fluticasone/Azelastine); Test type: Superiority; p = 0.003, Wilcoxon (Mann-Whitney); Median Difference (Net) = 4.5
Statistical Analysis 4: Comparison: Placebo vs Fluticasone Propionate; Test type: Superiority; p = 0.53, Wilcoxon (Mann-Whitney); Median Difference (Net) = 48.5

3. Other Pre Specified Outcome: Total Nasal Symptom Score
Description: Total nasal symptom Score = Sum of itchy, runny, sneezing, and congestion scores, each on scale 0-3 (0=no symptoms, 1=mild symptoms, 2=moderate symptoms, 3=severe symptoms). Thus, maximum=12, minimum=0, and higher score represents worse outcome. Measured in the 10 minute period after allergen challenge and normalized against symptoms experienced after sham challenge.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Fluticasone Propionate | Dymista (Fluticasone/Azelastine)
Number analyzed (Participants) | 19 | 19 | 19
score on a scale
  day 1 | 6.26 (0.85) | 7.06 (1.08) | 3.58 (0.81)
  day 2 | 6.63 (1.13) | 6.44 (0.91) | 4.32 (0.86)
  day 3 | 5.68 (1.07) | 5.67 (0.89) | 4.22 (0.88)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Propionate vs Dymista (Fluticasone/Azelastine); We used Friedman test to compare the distribution of total nasal symptom scores among three treatment groups (Placebo, Fluticasone propionate, Dymista) in each of the three days (day 1, day 2, and day 3); Test type: Superiority; p = 0.07, Friedman's Test — Alpha=0.05/3 since 3 days are compared; Friedman's Q = 5.22

4. Other Pre Specified Outcome: Change From Baseline Response in Lactoferrin Levels in Nasal Lavage Following Each Challenge
Description: Our procedure used a diluent (sham) challenge followed by 2 allergen challenges where lavages are collected 10 minutes after each of these challenges. The final value is (lactoferrin amount in lavage after 1st allergen exposure - amount after sham) + (amount in lavage after 2nd exposure - sham amount).
Time Frame: as for outcome 1
Population: There was one missing sample
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Fluticasone Propionate | Dymista (Fluticasone/Azelastine)
Number analyzed (Participants) | 18 | 18 | 18
ng/mL | 131368 (67483) | 137539 (40363) | 31400 (44982)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Propionate vs Dymista (Fluticasone/Azelastine); Test type: Superiority; p = 0.08, Friedman's Test — Bonferroni correction was used to adjust for the fact that each day was tested separately, giving alpha=0.05/3; Friedman's Q = 5.06

5. Other Pre Specified Outcome: Eosinophils
Description: Our procedure used a diluent (sham) challenge followed by 2 allergen challenges where lavages are collected 10 minutes after each of these challenges. The final value is (number of eosinophils in lavage after 1st allergen exposure - number after sham) + (number in lavage after 2nd exposure - sham number).
Time Frame: as for outcome 1
Population: due technical difficulty in the staining, no data is available.
Arm/Group | Placebo | Fluticasone Propionate | Dymista (Fluticasone/Azelastine)
Number analyzed (Participants) | 0 | 0 | 0

6. Other Pre Specified Outcome: Histamine
Description: Our procedure used a diluent (sham) challenge followed by 2 allergen challenges where lavages are collected 10 minutes after each of these challenges. The final value is (histamine amount in lavage after 1st allergen exposure - amount after sham) + (amount in lavage after 2nd exposure - sham amount).
Time Frame: as for outcome 1
Population: there were three missing samples
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Fluticasone Propionate | Dymista (Fluticasone/Azelastine)
Number analyzed (Participants) | 16 | 16 | 16
ng/mL | -0.97 (1.2) | 10.3 (7.6) | 12.3 (9.8)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Propionate vs Dymista (Fluticasone/Azelastine); Test type: Superiority; p = 0.04, Friedman's Test — Bonferroni correction was used to adjust for the fact that each day was tested separately, giving alpha=0.05/3; Friedman's Q = 6.53

7. Other Pre Specified Outcome: Tryptase
Description: Our procedure used a diluent (sham) challenge followed by 2 allergen challenges where lavages are collected 10 minutes after each of these challenges. The final value is (tryptase amount in lavage after 1st allergen exposure - amount after sham) + (amount in lavage after 2nd exposure - sham amount).
Time Frame: as for outcome 1
Population: Data was missing for 3 subjects
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Placebo | Fluticasone Propionate | Dymista (Fluticasone/Azelastine)
Number analyzed (Participants) | 16 | 16 | 16
ng/ml | -0.08 (0.28) | -0.19 (0.39) | 0.12 (0.26)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Propionate vs Dymista (Fluticasone/Azelastine); Test type: Superiority; p > 0.05, Friedman's Test — Bonferroni correction was used to adjust for the fact that each day was tested separately, giving alpha=0.05/3; Friedman's Q = 0.53

8. Other Pre Specified Outcome: Eosinophil Cationic Protein (ECP)
Description: Our procedure used a diluent (sham) challenge followed by 2 allergen challenges where lavages are collected 10 minutes after each of these challenges. The final value is (ECP amount in lavage after 1st allergen exposure - amount after sham) + (amount in lavage after 2nd exposure - sham amount).
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Fluticasone Propionate | Dymista (Fluticasone/Azelastine)
Number analyzed (Participants) | 19 | 19 | 19
ng/mL
  day 1 | 47.08 (14.67) | 47.8 (13.46) | 51.62 (13.03)
  day 2 | 44.5 (13.18) | 36.13 (11) | 46.32 (14.65)
  day 3 | 42.4 (10.25) | 37.91 (10.77) | 53.33 (16.14)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Propionate vs Dymista (Fluticasone/Azelastine); Test type: Superiority; p = 0.85, Friedman's Test — Bonferroni correction was used to adjust for the fact that each day was tested separately, giving alpha=0.05/3; Friedman's Q = 0.33

ADVERSE EVENTS:
Time Frame: with one month of patient study completion
Description: does not differ
Arm/Group | Placebo | Fluticasone Propionate | Dymista (Fluticasone/Azelastine)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-21): https://cdn.clinicaltrials.gov/large-docs/65/NCT02402465/Prot_SAP_000.pdf
  • Informed Consent Form (2017-08-08): https://cdn.clinicaltrials.gov/large-docs/65/NCT02402465/ICF_001.pdf